CLINICAL TRIAL: NCT00277524
Title: OMNI Study--Assessing Therapies in Medtronic Pacemaker, Defibrillator, and Cardiac Resynchronization Therapy Devices.
Acronym: OMNI
Status: Terminated | Type: Observational
Why Stopped: Ended follow-up after four years
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor
Other Study IDs: 601
Record Dates: First submitted 2006-01-12; First posted 2006-01-16 (Estimated); Results first posted 2013-08-28 (Estimated); Last update posted 2013-08-28 (Estimated); Status verified 2013-05

CONDITIONS: Tachycardia, Ventricular; Heart Failure, Congestive; Ventricular Fibrillation; Ventricular Dysfunction; Bradycardia
Keywords: Pacemaker; Defibrillator; Cardiac Resynchronization; Dysynchrony; Heart failure; Arrhythmia; Tachycardia; Bradycardia
MeSH Terms: conditions — Tachycardia, Ventricular; Heart Failure; Ventricular Fibrillation; Ventricular Dysfunction; Bradycardia; Arrhythmias, Cardiac; Tachycardia

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Overall: All patients enrolled in OMNI. Patient sub-groups include device type, history of atrial fibrillation (AF), history of investigate atrioventricular (AV) block, implant indication, and managed ventricular pacing (MVP) enabled.

SUMMARY:
The purpose of the OMNI study is to characterize therapy and diagnostic utilization in study participants implanted with study devices and to describe Implantable Cardioverter Defibrillator(ICD)therapy utilization for life threatening arrhythmias in primary and secondary prevention study participants. This study will assess therapies in Medtronic pacemaker, defibrillator, and cardiac resynchronization therapy devices.

The first therapy is for reducing unnecessary pacing in pacemaker patients. The second therapy provides pacing therapy in an attempt to stop fast or life threatening ventricular arrhythmias in lieu of delivering a defibrillation shock. The third therapy is a diagnostic measurement of a patient's fluid status and provides the physician information on the patient's heart failure status.

The study will also assess the time to a patient's first defibrillation shock and will verify that the shock was for a fast or life threatening ventricular rhythm.

DETAILED DESCRIPTION:
The OMNI results demonstrate the importance of Medtronic's ongoing efforts to increase adoption of evidence based shock-reduction programming strategies. Longer VF NID (number of intervals to detect in the VF zone) should be utilized with the Anti-tachycardia Pacing (ATP) During Charging Feature. ATP during Charging allows physicians to treat with ATP without delay to shock. Therefore, VF NID may be extended to allow episodes the chance to self-terminate immediately to shock by use of the ATP during the charging feature.

ELIGIBILITY:
Inclusion Criteria:

* Implant of new or replacement study device. Enrollment must occur no later than 40 days post-implant.
* Study participants must be 18 years of age or older.

Exclusion Criteria:

* Study participants enrolled or intend to participate in another clinical device trial during the course of this study that required specific treatment or programming.
* Study participants unwilling and unable to comply with follow-up schedule.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients receiving a specified Medtronic Implantable Pulse Generator(IPG), Implantable Cardioverter Defibrillator(ICD), or Cardiac Resynchronization Therapy-Defibrillator(CRT-D) device where informed consent and/or authorization to use and disclose health information permission has been granted.
Sampling Method: Non-Probability Sample
Enrollment: 3032 (Actual)
Dates: Start 2005-08; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael O. Sweeney, Principal Investigator — Cardiovascular Division Brigham and Womens
Locations (113):
- United States (113):
  - Southern Arizona Health Care System, Tucson, Arizona
  - Arkansas Cardiology PA (Little Rock AR), Little Rock, Arkansas
  - California Heart Medical Associates, Fresno, California
  - Apex Cardiology, Inglewood, California
  - Scripps Green Hospital Scripps Clinic Torrey Pines, La Jolla, California
  - Northern California Heart Care, Larkspur, California
  - Mission Internal Medical Group, Mission Viejo, California
  - Orange County Heart Institute & Research Center, Orange, California
  - Foothill Cardiology, Pasadena, California
  - Desert Cardiology Center / Desert Cardiology Medical Group Consultants, Rancho Mirage, California
  - Brett Berman Cardiology & Cardiac Electrophysiology, San Diego, California
  - Dwain L Coggins MD FACC, San Jose, California
  - Cardiology Clinic of San Antonio, Tarzana, California
  - Erol Kosar MD Inc, Torrance, California
  - Rocky Mountain Cardiology PC, Boulder, Colorado
  - Pikes Peak Cardiology, Colorado Springs, Colorado
  - Daytona Heart, Daytona Beach, Florida
  - Florida Arrhythmia Consultants, Fort Lauderdale, Florida
  - Clark & Daughtrey Medical Group PA, Lakeland, Florida
  - Melbourne Internal Medicine Associates / Century Research Associates, Melbourne, Florida
  - C. Raghavan MD PA, Orlando, Florida
  - Northwest Florida Heart Group PA, Pensacola, Florida
  - Heart & Vascular Institute of Florida, Safety Harbor, Florida
  - Florida Cardiovascular Institute PA, Tampa, Florida
  - Interventional Cardiac Consultants PLC, Trinity, Florida
  - Emory University Hospital, Atlanta, Georgia
  - Northeast Georgia Heart Center PC, Gainesville, Georgia
  - Macon Electrophysiology Associates PC, Macon, Georgia
  - Cardiovascular Consultants (Savannah GA), Savannah, Georgia
  - Edward N Shen MD Inc, Honolulu, Hawaii
  - Midwest Cardiology PC, Belleville, Illinois
  - Cardiovascular Associates, Elk Grove Village, Illinois
  - The Heart Group PC, Evansville, Indiana
  - Saint Mary Medical Center (Community Healthcare System), Hobart, Indiana
  - Cardiologists PC, Cedar Rapids, Iowa
  - King's Daughters Medical Center, Ashland, Kentucky
  - University Medical Associates, Louisville, Kentucky
  - Cardiovascular Associates LLC, Covington, Louisiana
  - Cardiology Associates PC, Annapolis, Maryland
  - Cardiovascular Specialists of Frederick, Frederick, Maryland
  - The Heart Center, Glen Burnie, Maryland
  - Baltimore Heart Associates (Randallstown MD), Randallstown, Maryland
  - Shady Grove Adventist Hospital, Rockville, Maryland
  - Peninsula Cardiology Associates, Salisbury, Maryland
  - Internal Medicine & Cardiology Associates of Southeastern New England PC, Fall River, Massachusetts
  - New Bedford Medical Associates, New Bedford, Massachusetts
  - North Shore Cardiology Associates, Salem, Massachusetts
  - University of Massachusetts Memorial Medical Center, Worcester, Massachusetts
  - University of Michigan Health System (UMHS) VA Medical Center, Ann Arbor, Michigan
  - Genesys Regional Medical Center, Grand Blanc, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - Cardiology Consultants of East Michigan, Lapeer, Michigan
  - Great Lakes Heart and Vascular Institute PC, Saint Joseph, Michigan
  - Cardiovascular Clinical Associates PC, Southfield, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Saint Paul Cardiology, Saint Paul, Minnesota
  - Hattiesburg Clinic/Forrest General, Hattiesburg, Mississippi
  - Cardiovascular Consultants (Cape Giradeau MO), Cape Girardeau, Missouri
  - Cardiology Consultants of Saint Louis County PC, St Louis, Missouri
  - Saint Louis Heart & Vascular PC, St Louis, Missouri
  - Heart Consultants PC, Omaha, Nebraska
  - Reno Heart Physicians, Reno, Nevada
  - New Jersey Heart (Elizabeth NJ), Elizabeth, New Jersey
  - Englewood Hospital & Medical Center, Englewood, New Jersey
  - Saint Joseph's Regional Medical Center, Paterson, New Jersey
  - Cardiology Associates, Woodland Park, New Jersey
  - Albany Associates in Cardiology, Albany, New York
  - Cardio Research of New York Inc, Bayside, New York
  - New York Medical Center of Queens, New York, New York
  - Heartwise Cardiology, New York, New York
  - Arrhythmia Associates of New York, New York, New York
  - University Cardiovascular Associates (UCVA), Rochester, New York
  - Cardiology Associates of Schenectady PC, Schenectady, New York
  - Saint Catherine of Sienna Medical Center, Smithtown, New York
  - Sanger Heart and Vascular Institute-Charlotte, Charlotte, North Carolina
  - Heart Rhythm Associates PLLC, Greenville, North Carolina
  - High Point Regional Health System, High Point, North Carolina
  - Wake Heart & Vascular Associates, Raleigh, North Carolina
  - Wilmington Cardiology LLC, Wilmington, North Carolina
  - Forsyth Medical Center, Winston-Salem, North Carolina
  - Altru Hospital, Grand Forks, North Dakota
  - TriHealth Good Samaritan Hos, Cincinnati, Ohio
  - EMH Elyria Medical Center, Elyria, Ohio
  - Heart Care Inc, Gahanna, Ohio
  - Stark Medical Specialties Inc, Massillon, Ohio
  - Ohio Institute of Cardiac Care Inc, Springfield, Ohio
  - The Toledo Clinic, Toledo, Ohio
  - Bluestem Cardiology PC, Bartlesville, Oklahoma
  - Heart Consultants, Midwest City, Oklahoma
  - Terrance Khastgir MD PC, Oklahoma City, Oklahoma
  - Pacific Heart Associates, Portland, Oregon
  - Altoona Regional Health Center, Altoona, Pennsylvania
  - Arrhythmia Institute, Newtown, Pennsylvania
  - Cardiology Consultants of Philadelphia, Philadelphia, Pennsylvania
  - Marshall-Rismiller & Associates, Pottsville, Pennsylvania
  - Columbia Heart Clinic PA, Columbia, South Carolina
  - Pee Dee Cardiology, Florence, South Carolina
  - Piedmont Cardiology Associates (Greenwood SC), Greenwood, South Carolina
  - Memphis Heart Clinic, Memphis, Tennessee
  - James H Quillen VA Medical Center, Mountain Home, Tennessee
  - Amarillo Heart Group, Amarillo, Texas
  - Dallas VA Medical Center, Dallas, Texas
  - Hall Garcia Cardiology Associates, Houston, Texas
  - Heart Clinic PLLC, McAllen, Texas
  - Medical Center Hospital Odessa, Odessa, Texas
  - Cardiology Clinic of San Antonio, San Antonio, Texas
  - Cardiovascular Associates of East Texas PA, Tyler, Texas
  - Utah Cardiology (Ogden UT), Ogden, Utah
  - Virginia Cardiovascular Specialists PC, Richmond, Virginia
  - CAMC Institute Clinical Trials Center, Charleston, West Virginia
  - Wisconsin Heart SC, Madison, Wisconsin
  - Arrhythmia Consultants of Milwaukee SC, Wauwatosa, Wisconsin

REFERENCES:
- [Background] Wathen MS, DeGroot PJ, Sweeney MO, Stark AJ, Otterness MF, Adkisson WO, Canby RC, Khalighi K, Machado C, Rubenstein DS, Volosin KJ; PainFREE Rx II Investigators. Prospective randomized multicenter trial of empirical antitachycardia pacing versus shocks for spontaneous rapid ventricular tachycardia in patients with implantable cardioverter-defibrillators: Pacing Fast Ventricular Tachycardia Reduces Shock Therapies (PainFREE Rx II) trial results. Circulation. 2004 Oct 26;110(17):2591-6. doi: 10.1161/01.CIR.0000145610.64014.E4. Epub 2004 Oct 18. PMID 15492306
- [Background] Alpert JS. Are data from clinical registries of any value? Eur Heart J. 2000 Sep;21(17):1399-401. doi: 10.1053/euhj.2000.2265. No abstract available. PMID 10952831
- [Background] Lamas GA, Williams A. Have the results of randomized clinical trials of pacing altered the practice of cardiac pacing? J Cardiovasc Electrophysiol. 2003 Sep;14(9 Suppl):S15-9. doi: 10.1046/j.1540-8167.14.s9.14.x. PMID 12950512
- [Background] Bardy GH, Lee KL, Mark DB, Poole JE, Packer DL, Boineau R, Domanski M, Troutman C, Anderson J, Johnson G, McNulty SE, Clapp-Channing N, Davidson-Ray LD, Fraulo ES, Fishbein DP, Luceri RM, Ip JH; Sudden Cardiac Death in Heart Failure Trial (SCD-HeFT) Investigators. Amiodarone or an implantable cardioverter-defibrillator for congestive heart failure. N Engl J Med. 2005 Jan 20;352(3):225-37. doi: 10.1056/NEJMoa043399. PMID 15659722
- [Background] Liang KY, Zeger S. Longitudinal data analysis using generalized linear models. Biometrika, 1986, 73:13-22.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study included 147 outpatient cardiology practices in the United States. Inclusion criteria were(1) implant of an implantable pulse generator (IPG), implantable cardioverter defibrillator (ICD) or cardiac resynchronization therapy defibrillator (CRT-D); and (2) age 18 years or older. Enrollment period was from Aug 2005 to Jun 2006.
Pre-assignment Details: This is a post-market prospective study. No group assignment is given. Subjects implanted with IPGs were enrolled and followed at 6 and 12 months. Subjects implanted with ICDs or CRT-Ds were enrolled and followed at six, 12, 24, 36, 48, and 60 months.
Groups:
- Subjects With IPG: Subjects implanted with an implantable pulse generator (IPG).
- Subjects With Single Chamber ICD: Subjects implanted with a single chamber implantable cardioverter defibrillator (ICD).
- Subjects With Dual Chamber ICD: Subjects implanted with a dual chamber implantable cardioverter defibrillator (ICD).
- Subjects With CRT-D: Subjects implanted with a cardiac resynchronization therapy defibrillator (CRT-D).
Period: Overall Study
Arm/Group | Subjects With IPG | Subjects With Single Chamber ICD | Subjects With Dual Chamber ICD | Subjects With CRT-D
Started | 621 | 324 | 1088 | 850
Completed | 621 | 324 | 1088 | 850
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Subjects implanted with an IPG, ICD or CRT-D and age 18 years or older were eligible for the OMNI study. Clinical data and device programming at baseline from all subjects was summarized for categorical and continuous variables using descriptive statistics.
Groups:
- Overall: All patients enrolled in OMNI.
Arm/Group | Overall
Number analyzed (Participants) | 2883
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 988
  >=65 years | 1895
Age Continuous [Mean (Standard Deviation); unit: years] | 68.7 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 907
  Male | 1976
Race/Ethnicity, Customized [Number; unit: participants] — 2817 subjects had information on race or ethnic origin.
  participants
    American Indian | 7
    Asian | 38
    Black | 335
    Hispanic | 206
    Native Hawaiian | 8
    White | 2217
    Other | 6
Region of Enrollment [Number; unit: participants]
  United States | 2883
Weight [Mean (Standard Deviation); unit: lbs] — 2781 subjects had information on weight.
  lbs | 188 (45.3)
QRS duration [Mean (Standard Deviation); unit: ms] — 2132 subjects had information on QRS duration.
  ms | 119.9 (34.0)
PR interval [Mean (Standard Deviation); unit: ms] — 1829 subjects had information on PR interval.
  ms | 182.6 (45.5)
LVEF(%) [Mean (Standard Deviation); unit: participants] — 2487 subjects had information on left ventricular ejection fraction (LVEF, %).
  participants | 33.4 (15.7)
New York Heart Association (NYHA) classification [Number; unit: participants] — New York Heart Association (NYHA) classification is used to classify the extent of heart failure. It has four classes: Class I (Mild), Class II (Mild), Class III (Moderate), and Class IV (Severe).
  participants
    I | 104
    II | 627
    III | 857
    IV | 72
    No Heart Failure | 600
    Missing | 5
Heart failure (HF) stage [Number; unit: participants] — This is a new classification heart failure (HF) which include four stages:
  Stage A - At high risk for HF but without structural heart disease or symptoms of HF; Stage B - Structural heart disease but without signs or symptoms of HF; Stage C - Structural heart disease with prior or current symptoms of HF; Stage D - Refractory HF requiring specialized interventions.
  participants
    A | 44
    B | 229
    C | 713
    D | 44
    No HF | 578
    NA | 1275
Number of patients implanted [Number; unit: participants] | 2882

OUTCOME MEASURES:

1. Primary Outcome: Implanted Systems Frequencies
Description: Frequencies of implanted systems were measured among patients who were implanted with a device (IPT, ICD or CRT-D).
Time Frame: Baseline
Measure: Number; unit: participants
Groups:
- Implanted Subjects: All patients enrolled in OMNI.
Arm/Group | Implanted Subjects
Number analyzed (Participants) | 2882
participants
  EnRhythm (P1501DR) | 620
  EnTrust AT (D154ATG) | 820
  EnTrust VR (D154VRC) | 321
  InSync Sentry (7297) | 30
  InSync Sentry (7299) | 820
  Intrinsic DR (7288) | 271

2. Primary Outcome: Implantable Pulse Generator (IPG) Device Baseline Programming Frequencies.
Description: Pacing mode is based on the NASPE/BPEG Generic (NBG) Pacemake coding which includes: I, the chambers paced (V= Ventricle, A=Atrium, D=Dual (A&V), O=None); II, the chambers sensed (V= Ventricle, A=Atrium, D=Dual (A&V), O=None); III, the mode of response (T=Triggered, I=Inhibited, D=Dual Triggered/Inhibited, O=None); IV, the programmable functions(R=Rate Modulated, C=Communicating, M=Multiprogrammable, P=Simple Programmable, O=None); V, the antitachycardia functions (O=None, P=Paced, S=Shocks, D=Dual (P&S)). In addition, MVP (managed ventricular pacing) is a mode that promotes AV conduction by reducing or eliminating unnecessary RV pacing but maintains dual chamber ventricular support in the event that AV conduction is lost.
Time Frame: Baseline
Measure: Number; unit: participants
Groups:
- IPG Group: Subjects implanted with IPG
Arm/Group | IPG Group
Number analyzed (Participants) | 620
participants
  Pacing Mode, DDD/DDDR | 81
  Pacing Mode, DDI/DDIR | 4
  Pacing Mode, MVP_AAIR_DD | 380
  Pacing Mode, MVP_AAI_DDD | 148
  Pacing Mode, VVI/VVIR | 7

3. Primary Outcome: ICD/CRT-D Device Baseline Programming Frequencies
Description: ICD/CRT-D baseline programming, pacing mode and detection. Pacing mode is based on the NASPE/BPEG Generic (NBG) Pacemake coding which includes: I, the chambers paced (V= Ventricle, A=Atrium, D=Dual (A&V), O=None); II, the chambers sensed (V= Ventricle, A=Atrium, D=Dual (A&V), O=None); III, the mode of response (T=Triggered, I=Inhibited, D=Dual Triggered/Inhibited, O=None); IV, the programmable functions(R=Rate Modulated, C=Communicating, M=Multiprogrammable, P=Simple Programmable, O=None); V, the antitachycardia functions (O=None, P=Paced, S=Shocks, D=Dual (P&S)). In addition, MVP (managed ventricular pacing) is a mode that promotes AV conduction by reducing or eliminating unnecessary RV pacing but maintains dual chamber ventricular support in the event that AV conduction is lost.
Time Frame: Baseline
Measure: Number; unit: participants
Units Other Than Participants: ICD/CRT-D Devices
Groups:
- ICD/CRT-D Group: Subjects implanted with ICD/CRT-D
Arm/Group | ICD/CRT-D Group
Number analyzed (Participants) | 2262
Number analyzed (ICD/CRT-D Devices) | 2262
participants
  Pacing Mode, DDD/DDDR | 804
  Pacing Mode, DDI/DDIR | 21
  Pacing Mode, MVP_AAIR_DD | 525
  Pacing Mode, MVP_AAI_DDD | 481
  Pacing Mode, VVI/VVIR | 424
  ATP Status, Before Charging | 23
  ATP Status, During Charging | 1089
  ATP Status, Off | 26
  VF Detection Enable, On | 2234
  VT Detection Enable, On | 1283
  VT Detection Enable, Monitor | 345
  VF Initial NID, 12/16 | 1176
  VF Initial NID, 18/24 | 1077
  VF Initial NID, 24/32 | 2
  FVT Detection On via VF zone | 829
  FVT Detection On via VT zone | 27

4. Secondary Outcome: AV Block Status by Device Type at 6 and 12 Months.
Description: Frequencies of subject with AV block over time between ICD and Implantable Pulse Generator(IPG) study participants.
Time Frame: 12 months post enrollment
Measure: Number; unit: participants
Groups:
- IPG (N=610): IPG Patients with MVP enabled and follow up data available
- ICD (N=1029): ICD Patients with MVP enabled and follow up data available
Arm/Group | IPG (N=610) | ICD (N=1029)
Number analyzed (Participants) | 610 | 1029
participants
  6 Months: Subjects with MVP enabled, N | 441 (12.5) | 815
  6 Months: AV Block 1st degree | 103 | 167
  6 Months: AV Block 2nd degree Type I | 11 | 7
  6 Months: AV Block 2nd degree Type II | 19 | 7
  6 Months: AV Block 3rd degree Intermittent | 39 | 5
  6 Months: AV Block 3rd degree Persistent | 11 | 5
  6 Months: None | 250 | 603
  12 Months: Subjects with MVP enabled, N | 389 | 732
  12 Months: AV Block 1st degree | 90 | 159
  12 Months: AV Block 2nd degree Type I | 12 | 7
  12 Months: AV Block 2nd degree Type II | 7 | 7
  12 Months: AV Block 3rd degree Intermittent | 30 | 5
  12 Months: AV Block 3rd degree Persistent | 14 | 7
  12 Months: None | 216 | 523

5. Secondary Outcome: AV Block Status by Severity of Historical AV Block
Description: Frequencies of Subjects with AV Block Over Time by Severity of Historical AV Block
Time Frame: 4 years post implant
Measure: Number; unit: participants
Groups:
- Patients Without History of AV Block; Patients With History of AV Block: Patients with MVP enabled and follow up data available
Arm/Group | Patients Without History of AV Block | Patients With History of AV Block
Number analyzed (Participants) | 1098 | 541
participants
  6 Months: Subjects with MVP enabled | 883 | 373
  6 Months: AV Block 1st degree | 49 | 221
  6 Months: AV Block 2nd degree Type I | 1 | 17
  6 Months: AV Block 2nd degree Type II | 1 | 25
  6 Months: AV Block 3rd degree Intermittent | 2 | 42
  6 Months: AV Block 3rd degree Persistent | 3 | 13
  6 Months: None | 818 | 35
  12 Months: Subjects with MVP enabled | 786 | 335
  12 Months: AV Block 1st degree | 73 | 176
  12 Months: AV Block 2nd degree Type I | 0 | 19
  12 Months: AV Block 2nd degree Type II | 1 | 13
  12 Months: AV Block 3rd degree Intermittent | 5 | 30
  12 Months: AV Block 3rd degree Persistent | 3 | 18
  12 Months: None | 689 | 50
  24 Months: Subjects with MVP enabled | 426 | 146
  24 Months: AV Block 1st degree | 51 | 95
  24 Months: AV Block 2nd degree Type I | 0 | 5
  24 Months: AV Block 2nd degree Type II | 0 | 3
  24 Months: AV Block 3rd degree Intermittent | 1 | 3
  24 Months: AV Block 3rd degree Persistent | 0 | 2
  24 Months: None | 362 | 24
  36 Months: Subjects with MVP enabled | 324 | 105
  36 Months: AV Block 1st degree | 58 | 69
  36 Months: AV Block 2nd degree Type I | 1 | 3
  36 Months: AV Block 2nd degree Type II | 0 | 2
  36 Months: AV Block 3rd degree Intermittent | 0 | 3
  36 Months: AV Block 3rd degree Persistent | 0 | 2
  36 Months: None | 253 | 18
  48 Months: Subjects with MVP enabled | 269 | 92
  48 Months: AV Block 1st degree | 59 | 59
  48 Months: AV Block 2nd degree Type I | 0 | 2
  48 Months: AV Block 2nd degree Type II | 0 | 1
  48 Months: AV Block 3rd degree Intermittent | 0 | 2
  48 Months: AV Block 3rd degree Persistent | 1 | 2
  48 Months: None | 201 | 17

6. Secondary Outcome: Summary of ATP Episodes Within All Treated Episodes
Description: Evaluate the utility of the Antitachycardia Pacing (ATP) During Charging feature of the device.
Time Frame: 4 years post enrollment
Measure: Number; unit: Episodes
Groups:
- ATP During Charging: Patients who had an episode and were programmed with the ATP during charging feature.
Arm/Group | ATP During Charging
Number analyzed (Participants) | 343
Episodes
  Number of episodes analyzed from 343 participants | 1584
  Episodes with ATP attempted | 1100
  Episodes with Sucessful ATP | 650

7. Secondary Outcome: Compare First Shock Rate Between Medtronic "PainFREE" Programming and "SCD-HeFT" Programming in Primary Prevention Study Participants.
Description: First shock rate for VF and FVT zones was estimated using Kaplan-Meier method.
  OMNI "PainFREE" definition: programming combinations that result in ATP therapy for ventricular tachycardia (VT) at cycle lengths <320 ms. Programming at cycle lengths ≥320 ms were not mandated.
  OMNI "SCD-HeFT" definition: programming combinations that result in shock therapy only for arrhythmias at cycle lengths of <320 ms or faster and no therapy for arrhythmias at cycle lengths ≥320 ms.
Time Frame: 4 years post implant
Measure: Mean (Standard Deviation); unit: rate
Groups:
- "PainFREE" Programming: OMNI "PainFREE" definition: programming combinations that result in ATP therapy for VT at cycle lengths <320 ms. Programming at cycle lengths ≥320 ms were not mandated.
- "SCD-HeFT" Programming: OMNI "SCD-HeFT" definition: programming combinations that result in shock therapy only for arrhythmias at cycle lengths of <320 ms or faster and no therapy for arrhythmias at cycle lengths ≥320 ms.
Arm/Group | "PainFREE" Programming | "SCD-HeFT" Programming
Number analyzed (Participants) | 1116 | 462
rate
  At implant | 0 (0) | 0 (0)
  12 months after implant | 0.10 (0.009) | 0.15 (0.017)
  24 months after implant | 0.14 (0.011) | 0.21 (0.019)
  36 months after implant | 0.18 (0.013) | 0.24 (0.021)
  48 months after implant | 0.20 (0.014) | 0.27 (0.023)

8. Secondary Outcome: Frequencies of Subjects With OptiVol Trends and Disease Progression.
Description: Estimate the correlation between OptiVol trends and disease progression.
  A subject's disease status was said to have progressed if:
  1. The NYHA classification number increases (example: I to II), or
  2. The LVEF decreases by at least 20% (relative difference) and by at least a 5% absolute difference, or
  3. The subject expires
  A subject who crossed OptiVol threshold since last visit was regarded as 'crossed threshold'.
Time Frame: 4 years post implant
Measure: Number; unit: participants
Groups:
- 12-month Follow-up: Total subjects with disease progressed at 12 months
- 24-month Follow-up: Total subjects with disease progressed at 24 months
- 36-month Follow-up: Total subjects with disease progressed at 36 months
- 48-month Follow-up: Total subjects with disease progressed at 48 months
Arm/Group | 12-month Follow-up | 24-month Follow-up | 36-month Follow-up | 48-month Follow-up
Number analyzed (Participants) | 488 | 375 | 326 | 257
participants
  Disease Progressed, N | 97 | 95 | 93 | 84
  Crossed Threshold, N | 382 | 327 | 287 | 224

9. Primary Outcome: ICD/CRT-D Device Baseline Programming Measurements
Description: ICD/CRT-D baseline programming measurements, detection interval. Implanted Cardioverter/Defibrillator paces a patient's heart in a tachyarrhythmia prevention-pacing mode.
  Detection intervals are used to detect atrial tachyarrhythmia. Detection Intervals are programmable heart rate thresholds. R-R intervals that are less than the VT or VF detection intervals (in ms) are considered evidence of VT or VF, respectively. R-R intervals that are between the FVT and the VF detection intervals are considered evidence of FVT. Thus, these detection interval thresholds demarcate rate zones of detection. The rate zones are used to determine the type of therapy applied once detection occurs.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: ms
Groups:
- ICD/CRT-D Group: Subjects implanted with Implantable Cardioverter Defibrillator, Cardiac Resynchronization Therapy-Defibrillator (ICD/CRT-D).
Arm/Group | ICD/CRT-D Group
Number analyzed (Participants) | 2262
ms
  Pace AV | 168 (39.2)
  Sense AV | 139 (40.8)
  FVT Detection Interval | 260 (24.6)
  VF Detection Interval | 314 (17.1)
  VT Detection Interval | 383 (25.2)

ADVERSE EVENTS:
Description: The Medtronic OMNI Study is a post-market observational study conducted in the United States (US). Adverse events were not collected as a part of the OMNI study. Sites were instructed to report applicable events in the same manner as required for any commercially available device, through the Medical Device Reporting (MDR) process.
Groups:
- EG000: The Medtronic OMNI Study is a post-market observational study conducted in the United States (US). Adverse events were not collected as a part of the OMNI study. Sites were instructed to report applicable events in the same manner as required for any commercially available device, through the Medical Device Reporting (MDR) process.
Arm/Group | EG000
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No